CLINICAL TRIAL: NCT02391909
Title: Phase 4 Observational Prospective Cohort Study to Assess the Safety of Vivotif at Different Release Titers Among Travelers
Brief Title: Phase 4 Study To Assess The Safety Of Vivotif At Different Release Titers Among Travelers
Status: Completed | Type: Observational
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: VIV-PASS-01
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Typhoid Fever
Keywords: Vaccine
MeSH Terms: conditions — Typhoid Fever | interventions — Ty21a typhoid vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Vivotif 6.9-10.0 x109 CFU/capsule
  Interventions: Biological: Vivotif
- Group B: Vivotif 4.0-6.8 x109 CFU/capsule
  Interventions: Biological: Vivotif

INTERVENTIONS:
Biological: Vivotif

SUMMARY:
This is a multicenter (at travel clinics), phase 4 observational prospective cohort study in healthy adult male and female travelers for whom typhoid vaccination with Vivotif is recommended, as per standard practice.

DETAILED DESCRIPTION:
This is a multicenter (at travel clinics), phase 4 observational prospective cohort study in healthy adult male and female travelers for whom typhoid vaccination with Vivotif is recommended, as per standard practice.

The study will enroll 950 subjects who will be randomized at a ratio of 1:1 into two groups, A and B, of 475 subjects each. Group A will receive 6.9-10.0 x109 CFU/capsule and Group B will receive 4.0-6.8 x109 CFU/capsule, respectively.

All subjects will receive four doses of Vivotif. One dose per subject will be administered on Days 1, 3, 5 and 7.

Investigators, subjects and all personnel involved in running the study will not be aware of the actual release titer associated with the distributed lots. Blinding is maintained using the commercial packaging that does not include the actual value of the release titer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are male or female aged ≥ 18 years at time of dosing
2. Subjects are travelers attending travelers' vaccination clinics
3. Subjects are eligible for typhoid vaccination, according to standard practice
4. Subjects are expected to be able to provide follow-up information
5. Subjects have an expected travel departure date more than 21 days after enrollment (to enhance follow-up by ensuring subjects remain in the US during the AE collection period)
6. Subjects must sign a written informed consent

Exclusion Criteria:

1. Subjects with a known hypersensitivity to any component of the vaccine or the enteric coated capsule
2. Subjects deficient in their ability to mount a humoral or cell-mediated immune response due to either a congenital or acquired immunodeficient state including treatment with immune-suppressive or antimitotic drugs
3. Subjects with an acute febrile illness
4. Subjects with acute gastrointestinal (GI) illness
5. Subjects who are receiving medications with antibacterial activity (including proguanil) at the time of enrollment
6. Subjects with other contraindications as determined by the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Travelers attending travelers' vaccination clinics, and for whom typhoid vaccination with Vivotif is recommended, according to standard practice
Sampling Method: Probability Sample
Enrollment: 855 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
The occurrence of any AE up to two weeks after the scheduled final vaccine dose | Day 21

SECONDARY OUTCOMES:
The distribution of the solicited Adverse Reactions | Day 21
The distribution of unsolicited Adverse Reactions | Day 21
The occurrence of any unsolicited adverse event up to two weeks after the scheduled final vaccine dose | Day 21
The occurrence of any SAE up to two weeks after the scheduled final vaccine dose | Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Passport Health, Baltimore, Maryland, United States